CLINICAL TRIAL: NCT01959997
Title: Randomized Comparison of Redo Pulmonary Vein Isolation With vs. Without Renal Denervation for Recurrent Atrial Fibrillation After Initial Pulmonary Vein Isolation
Brief Title: Comparison of Redo PVI With vs. Without Renal Denervation for Recurrent AF After Initial PVI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD_REDO_032
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation; Arterial Hypertension
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Redo PVI (Active Comparator): Therapeutic anticoagulation will be required for at least 3 weeks prior to ablation. An MRA will be performed to define cardiac and PV anatomy. Standard ablation technique will be employed. After gaining venous access, double transseptal puncture will be performed to permit left atrial access, guided by intracardiac ultrasound. A circular mapping catheter will be placed in each PV and any reconnections will be ablated by delivery of RF energy. Confirmation of re-isolation of all PVs will be performed at the conclusion of the procedure.
  Interventions: Procedure: Redo PVI
- PVI + RDN (Active Comparator): All patients who are randomized to Group II will undergo redo PVI exactly as described above.
  At the conclusion of PVI, RDN will be performed. Real-time 3-dimensional aorta-renal artery maps will be constructed with the use of the same navigation system and catheter used for PVI after femoral artery access. Both mapping and ablation will performed under the same modified sedation. RF ablations of 8 to 10 watts will be applied discretely from the first distal main renal artery bifurcation all the way back to the ostium, for 2 min, and up to 6 lesions (separated by ≥ 5 mm). Lesions will be made both longitudinally and rotationally within each renal artery. To confirm renal denervation, high-frequency stimulation (HFS) will be used before the initial and after each RF delivery within the renal artery. RDN will be considered to have been achieved when the sudden increase of blood pressure (≥ 15 mm Hg from invasive arterial monitoring) is absent.
  Interventions: Procedure: PVI + RDN

INTERVENTIONS:
Procedure: Redo PVI
  Arms: Redo PVI
Procedure: PVI + RDN
  Arms: PVI + RDN

SUMMARY:
The objective of this study is to compare the elimination of atrial fibrillation in patients with recurrent atrial fibrillation despite prior pulmonary vein isolation (PVI) when undergoing repeat PVI (control) vs repeat PVI plus renal denervation.

ELIGIBILITY:
Inclusion Criteria:

* Prior PVI ablation procedure for paroxysmal AF within past 2 years
* Recurrent symptomatic paroxysmal AF despite prior PVI
* History of essential hypertension requiring at least 2 chronic antihypertensive medications

Exclusion Criteria:

* Persistent AF after prior ablation
* Congestive heart failure (NYHA III-IV functional class)
* Left ventricle ejection fraction < 35%
* Left atrial diameter >55 mm
* An estimated glomerular filtration rate (eGFR) < 45mL/min/1.73m2, using the MDRD calculation
* Renal arteries unsuitable for RDN:

  1. Inability to access renal vasculature
  2. Main renal arteries < 4 mm in diameter or < 20 mm in length.
  3. Hemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery
  4. A history of prior renal artery intervention including balloon angioplasty or stenting that precludes a possibility of ablation treatment
  5. Multiple main renal arteries to either kidney
* Unwillingness to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The absence of AF | 1 year
  The absence of AF at one year as assessed by prolonged ambulatory ECG monitoring post-ablation after 3 month blanking period has expired following the repeat ablation procedure.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressures | 1 year
procedural duration and complications | 1 year
LV mass on echocardiogram | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S. Steinberg, MD, Principal Investigator — University of Rochester
Locations (2):
- University of Rochester, Rochester, New York, United States
- State Research Institute of Circulation Pathology, Novosibirsk, Russia